CLINICAL TRIAL: NCT06960018
Title: Controlled, Randomized Clinical Study to Demonstrate the Patient Benefit and Safety of Pedicle Screw Placement Through an Innovative Minimally Invasive Surgical Approach Using the Ennovate® Cervical Spinal System
Brief Title: Clinical Study on the Safety and Efficacy of the Minimally Invasive Ennovate® Method for Pedicle Screw Placement
Acronym: MISPEC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aesculap AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AAG-O-H-23045
Record Dates: First submitted 2025-04-16; First posted 2025-05-07 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Cervical Spine Disease; Pain, Postoperative
Keywords: posterior cervical fusion; pedicle screw
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: Subjects will be randomly allocated to one of the two study groups in a 1:1 ratio.
  In addition, stratification by clinical investigation sites is applied. Group 1: Patients treated with the Ennovate® Cervical system using an open surgical technique. Group 2: Patients treated with the Ennovate® Cervical system using a minimally invasive technique. Study is designed to provide a comparison of the both groups regarding the short-term pain outcome.
Who Masked: Participant
Masking Description: Block randomization with random block length will be used. The electronic data capture system will instruct the clinical investigator to use either the open or the minimally invasive surgical technique.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Implantation Ennovate® Cervical system using an open surgical technique (Active Comparator)
  Interventions: Device: Ennovate® Cervical, open surgical technique
- Implantation Ennovate® Cervical system using a minimally invasive technique. (Experimental)
  Interventions: Device: Ennovate® Cervical, minimal invasive surgical technique

INTERVENTIONS:
Device: Ennovate® Cervical, open surgical technique — Patients with need of posterior monosegmental and multisegmenta stabilization of the cervical and upper thoracic spine, because of
  * Fractures
  * Degenerative instability
  * Post-trauma instability
  * Tumors
  * Degenerative cervical myelopathy due to multilevel subaxial spinal canal stenosis will be treated with Ennovate® Cervical system using an open surgical technique
  Arms: Implantation Ennovate® Cervical system using an open surgical technique
Device: Ennovate® Cervical, minimal invasive surgical technique — Patients with need of posterior monosegmental and multisegmenta stabilization of the cervical and upper thoracic spine, because of
  * Fractures
  * Degenerative instability
  * Post-trauma instability
  * Tumors
  * Degenerative cervical myelopathy due to multilevel subaxial spinal canal stenosis will be treated with Ennovate® Cervical system using a minimally invasive technique.
  Arms: Implantation Ennovate® Cervical system using a minimally invasive technique.

SUMMARY:
The study's main purpose is the collection of clinical data on the patients benefit and safety of pedicle screw placement through an innovative minimally invasive surgical approach compared to the state of the art open surgical approach using the Ennovate® Cervical Spinal System.

ELIGIBILITY:
Inclusion Criteria:

* All patients with minimum 18 years of age receiving Ennovate® Cervical internal fixation device within the vertebral bodies C2-Th3 to ensure the restoration and stabilization of the cervical spine

Exclusion Criteria:

* All patients not willing to sign the patient consent are excluded. Also, if it is clear from the beginning, that the patient will not be able to come to routine follow-up, the patient will also be excluded.

Absolute contraindications according to the IFU:

* Severe damage to the bone structures of the spine that could prevent the stable implantation of the implant components; for example, osteopenia, severe osteoporosis, Paget's disease, bone tumors etc.
* Metabolic or degenerative metabolic bone diseases that could compromise the stable anchoring of the implant system.
* Suspected allergy or sensitivity to the implant materials.
* Acute or chronic vertebral infections of a local or systemic nature.
* Poor patient compliance or limited ability to follow medical instructions, particularly in the postop phase, including with regard to the restrictions on range of movement in terms of physical exercise and occupational activity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2025-06-20 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS) | 4 (+/- 1 day) postoperative
  Visual Analogue Scale (VAS) which state "0" at one end representing "no pain" and "100" at the opposite end representing "maximal/worst pain". Pain will be recorded at minimum 12 months postoperatively, if available in the preoperative clinical routine data, it will also be recorded in the study.

SECONDARY OUTCOMES:
Screw placement accuracy | intraoperative or discharge visit (approx. 10 days post op.)
  Evaluation of the accuracy of screw placement will be performed according to the method described by Bredow using CT/3D-Scans made at intraoperative/discharge visit.
Neck Disability Index (NDI) | praeoperative, postoperative (4 days +/- 1day, 2 weeks, 4 weeks, 6 weeks, 3 months, 1 year, 2 years)
  The Neck Disability Index (NDI) is a widely used and validated self-assessment tool for measuring disability due to neck pain. (Measured over the course of the study)
  * 0-4 (0-8%): No disability
  * 5-14 (10-28%): Mild disability
  * 15-24 (30-48%): Moderate disability
  * 25-34 (50-64%): Severe disability
  * 35-50 (70-100%): Complete disability
Quality of Life (EQ-5D-5L) | praeoperative, postoperative (4 days +/- 1day, 2 weeks, 4 weeks, 6 weeks, 3 months, 1 year, 2 years)
  EQ-5D is a standardized 5-dimension (5D) 5-level (5L) measure of the health status and is developed by the EuroQol Group in order to have a simple and generic measure for clinical and economic assessment. Instructions for the user are directly included into the questionnaire and it consists of two pages. One cover five different dimensions (mobility, self care, usual activities, pain/discomfort, anxiety/depression) and the other one the EQ visual Analogue Scale (EQ-VAS). The VAS scale records the self rated health status of the patient from the level "the worst health you can imagine" to "the best health you can imagine".
Quality of Life (EQ-VAS) | praeoperative, postoperative (4 days +/- 1day, 2 weeks, 4 weeks, 6 weeks, 3 months, 1 year, 2 years)
  EQ-5D is a standardized 5-dimension (5D) 5-level (5L) measure of the health status and is developed by the EuroQol Group in order to have a simple and generic measure for clinical and economic assessment. Instructions for the user are directly included into the questionnaire and it consists of two pages. One cover five different dimensions (mobility, self care, usual activities, pain/discomfort, anxiety/depression) and the other one the EQ visual Analogue Scale (EQ-VAS). The VAS scale records the self rated health status of the patient from the level "the worst health you can imagine" to "the best health you can imagine".
Rate of Adverse Events / Serious Adverse Events | During the course of the study up to two years postoperatively
  (Serious) Adverse Events During the course of the study, any upcoming intra- or postoperative (serious) adverse device events or effects ((S)AE) related or not related to the product under investigation, will be documented. The total number of (S)AEs will be summarized and further evaluated by the sponsor and reported according to local legislation and necessity. Recorded complications will be categorized and analyzed in order to assess the safety of the investigational product.
Visual Analogue Scale (VAS) | praeoperative, postoperative (2 weeks, 4 weeks, 6 weeks, 3 months, 1 year, 2 years)
  Visual Analogue Scale (VAS) which state "0" at one end representing "no pain" and "100" at the opposite end representing "maximal/worst pain". Pain will be recorded at minimum 12 months postoperatively, if available in the preoperative clinical routine data, it will also be recorded in the study.

CONTACTS AND LOCATIONS:
Locations (3):
- Germany (3):
  - Universitätsklinikum Aachen, Aachen
  - Charité Berlin, Berlin
  - Universitätsklinikum Freiburg, Freiburg im Breisgau

IPD SHARING:
Plan to Share IPD: No